CLINICAL TRIAL: NCT01775111
Title: Influence of Strength Training and Nutritional Supplementation on Physical Performance and Well-being of Older People in Pensioner Homes
Brief Title: Influence of Strength Training and Protein Supplementation on Fitness of Institutionalized Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Vienna (Other)
Collaborators: Kaiser Franz Josef Hospital (Other)
Responsible Party: Principal Investigator, Ass.-Prof. DI Dr. Barbara Wessner, Ass.Prof. DI Dr., University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ActiveAgeing
Record Dates: First submitted 2013-01-21; First posted 2013-01-24 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Aging
Keywords: strength training; protein supplementation; sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Cognitive Training; Resistance Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cognitive Training (Sham Comparator): Cognitive Training (riddles, skill games, ...) is performed twice a week in small groups
  Interventions: Behavioral: Cognitive Training
- Strength Training (Experimental): Progressive strength training is applied, meaning that the intensity is adjusted continuously in order to obtain a sufficient training stimulus. Exercises are chosen to involve the major muscle groups and are performed by using the own body weight or elastic bands.
  Interventions: Behavioral: Strength Training
- Strength Training and Supplement (Experimental): In addition to strength training as described above, participants receive a water-soluble dietary supplement 9x/week (FortiFit, Nutricia) consisting of 20.7 g of protein (56 En%, 19.7 g whey protein, 3 g leucine,> 10 g essential amino acids), 9.3 g carbohydrates (25 En%, 0.8 BE), 3.0 g fat (18 En%), 1.2 g fiber (2 En%), 800 IU (20μg) of vitamin D, 250mg calcium, vitamins B6 and B12, folic acid and magnesium.
  Interventions: Behavioral: Strength Training; Dietary Supplement: FortiFit

INTERVENTIONS:
Behavioral: Cognitive Training
  Arms: Cognitive Training
Behavioral: Strength Training
  Arms: Strength Training; Strength Training and Supplement
Dietary Supplement: FortiFit
  Arms: Strength Training and Supplement

SUMMARY:
The aim of this randomized, observer-blind, controlled intervention study with parallel groups is to study the effect of strength training (2x/week for 6 months) with and without additional dietary supplementation (protein-enriched) on muscle strength, function and mass, oxidative stress parameters and the immune system in elderly institutionalized persons.

The participants (n = 120) are recruited from Viennese senior residencies (Kuratorium Wiener Pensionistenwohnheime). After a pre-participation screening participants will be distributed randomly but stratified by sex and age to one of the 3 intervention groups (cognitive training, strength training, strength training + supplement).

Study participants are eligible if they are male or female with an age over 65 years and if their cognitive status as well as their physical fitness level allows to participate at the strength training sessions. Exclusion criteria comprise chronic diseases which contraindicate the medical training therapy, serious cardiovascular disease, diabetic retinopathy and manifest osteoporosis, medication with anticoagulants or cortisone drugs and also regular strength training during the last six months.

Primary outcome measure is the change in isokinetic torque of knee extensors. Secondary outcome measures comprise anthropometric data, functional performance tests, immunological and oxidative stress parameters. The change in muscle signaling pathways will be assessed from muscle biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Adequate mental condition in order to follow the instructions and to perform the resistance exercise independently (Mini-Mental-State >23)
* Ability to walk 10 meters independently (without orthopaedic devices)
* 4 or more points at the Short Physical Performance Battery

Exclusion Criteria:

* Chronic diseases, which contraindicate a medical training therapy
* Serious cardiovascular diseases (congestive chronic heart failure, severe or symptomatic aortic stenosis, unstable angina pectoris, untreated arterial hypertension, cardiac arrhythmias)
* Diabetic retinopathy
* Manifest osteoporosis
* Regular use of cortisone-containing drugs
* Regular strength training (> 1x / week) in the last 6 months before inclusion

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
change from baseline in isokinetic torque of knee extensors | baseline and 6 months

SECONDARY OUTCOMES:
change from baseline in 6min walking test | baseline and 6 months
change from baseline in handgrip strength | baseline and 6 months
change from baseline in single leg balance stand | baseline and 6 months
change from baseline in lean body mass | baseline and 6 months
change from baseline in muscular myostatin expression | baseline and 6 months
change from baseline in DNA strand breaks | baseline and 6 months
change from baseline in high-sensitive C reactive protein | baseline and 6 months

OTHER OUTCOMES:
change from baseline in isokinetic torque of knee extensors at 12 months | baseline and 12 months
change from baseline in isokinetic torque of knee extensors at 18 months | baseline and 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Wessner, Ass.-Prof. DI Dr., Principal Investigator — University of Vienna
Locations (1):
- University of Vienna, Centre of Sports Science and University Sports, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Franzke B, Schober-Halper B, Hofmann M, Oesen S, Tosevska A, Henriksen T, Poulsen HE, Strasser EM, Wessner B, Wagner KH. Age and the effect of exercise, nutrition and cognitive training on oxidative stress - The Vienna Active Aging Study (VAAS), a randomized controlled trial. Free Radic Biol Med. 2018 Jun;121:69-77. doi: 10.1016/j.freeradbiomed.2018.04.565. Epub 2018 Apr 24. PMID 29698742
- [Derived] Tosevska A, Franzke B, Hofmann M, Vierheilig I, Schober-Halper B, Oesen S, Neubauer O, Wessner B, Wagner KH. Circulating cell-free DNA, telomere length and bilirubin in the Vienna Active Ageing Study: exploratory analysis of a randomized, controlled trial. Sci Rep. 2016 Dec 1;6:38084. doi: 10.1038/srep38084. PMID 27905522
- [Derived] Grimpampi E, Oesen S, Halper B, Hofmann M, Wessner B, Mazza C. Reliability of gait variability assessment in older individuals during a six-minute walk test. J Biomech. 2015 Nov 26;48(15):4185-4189. doi: 10.1016/j.jbiomech.2015.10.008. Epub 2015 Oct 20. PMID 26515246